CLINICAL TRIAL: NCT00171652
Title: Efficacy and Safety of Diclofenac Sodium Gel in Hand Osteoarthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VOSG-PE-314
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2006-10-11 (Estimated); Status verified 2006-10

CONDITIONS: Osteoarthritis
Keywords: Hand osteoarthritis, Topical NSAID, Diclofenac sodium
MeSH Terms: conditions — Osteoarthritis

INTERVENTIONS:
Drug: Diclofenac sodium gel 1%

SUMMARY:
This study will test the efficacy and safety of topical diclofenac sodium gel in the treatment of hand osteoarthritis.

ELIGIBILITY:
Key Inclusion criteria:

• Osteoarthritis of the hand

Key Exclusion Criteria:

* Other rheumatic disease, such as rheumatoid arthritis
* Active gastrointestinal ulcer during the last year
* Known allergy to analgesic drugs

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360
Dates: Start 2005-05; Study Completion 2005-10

PRIMARY OUTCOMES:
OA pain intensity in target hand at Week 4 and 6
Total AUSCAN score in target hand at Week 4 and 6
Global rating of disease activity by patient at Week 4 and 6

SECONDARY OUTCOMES:
OA pain intensity and total AUSCAN score in target hand, and global rating of disease activity by patient at Weeks 1, 2 and 8
AUSCAN pain, stiffness and physical function scores in target hand, and global rating of benefit by patient at Weeks 1, 2, 4, 6 and 8
OA pain intensity in target hand and use of rescue medication recorded in diary
Global evaluation of treatment at final visit
Treatment responder rate according to OARSI criteria

CONTACTS AND LOCATIONS:
Locations (33):
- France (14):
  - Cergy
  - Clamart
  - Cournonterral
  - Fellering
  - Goussonville
  - Linas
  - Longpont-sur-Orge
  - Meaux
  - Nantes
  - Orly
  - Paris
  - Savigny-sur-Orge
  - Thouars
  - Villeneuve-le-Roi
- Germany (19):
  - Bad Hersfeld
  - Bad Nauheim
  - Berlin
  - Bochum
  - Dinslaken
  - Dortmund
  - Dreieich
  - Dresden
  - Frankfurt a/M
  - Hagen
  - Hamburg
  - Karlsruhe
  - Kassel
  - Leipzig
  - Ludwigshafen
  - München
  - Neustadt/Aisch
  - Nuremberg
  - Stuttgart

REFERENCES:
- [Derived] Barthel HR, Peniston JH, Clark MB, Gold MS, Altman RD. Correlation of pain relief with physical function in hand osteoarthritis: randomized controlled trial post hoc analysis. Arthritis Res Ther. 2010;12(1):R7. doi: 10.1186/ar2906. Epub 2010 Jan 11. PMID 20064249